CLINICAL TRIAL: NCT03923062
Title: Different Dermatological Approaches in Treatment of Melasma: A Split Face Randomized Clinical Trial
Brief Title: Different Dermatological Approaches the Treatment of Melasma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Hafez, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DDATM
Record Dates: First submitted 2019-04-01; First posted 2019-04-22 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G I A (right side): will be treated by chemical peeling (Experimental): right sideof patient's face will be treated by chemical peeling( Trichloroacetic acid 20% concentration).
  Interventions: Device: chemicalpeeling
- G I B(left side):will be treated by cryopeeling (Experimental): left side of the patient's face will be treated by cryopeeling using Liquid Nitrogen.
  Interventions: Device: cryopeeling
- G II A (right side): will be treated by chemical peeling (Experimental): right sideof patient's face will be treated by chemical peeling( Trichloroacetic acid 20% concentration).
  Interventions: Device: chemicalpeeling
- G II B (left side):will be treated by tranexemic acid (Experimental): left side of patient's face will be treated by tranexemic acid(cyclokapron)
  Interventions: Combination Product: microneedling

INTERVENTIONS:
Device: chemicalpeeling — Cleansing and degreasing the face with alcohol .
  * The patients must be sitting at an angle of 45.
  * A 2 × 2 cm cotton gauze will be used to apply TCA 20%.
  * We will apply the acid from the midline to the right side of the forehead and under the right eye, covering the right cheek and perioral area.
  * We then will wait for a few minutes and will observe the frost developing.
  * The patient will be then allowed to wash her face.
  Other Names: chemical peeling using Trichloroacetic acid 20%
  Arms: G I A (right side): will be treated by chemical peeling; G II A (right side): will be treated by chemical peeling
Device: cryopeeling — Cryopeeling will be performed by spraying the freezing substance(Liquid Nitrogen) on the face at 1-2cm distance and moving along the affected area until freezing appear.
  Other Names: cryopeeling using Liquid Nitrogen
  Arms: G I B(left side):will be treated by cryopeeling
Combination Product: microneedling — Tranexamic acid will be used in aconcentration of 4mg/ml ,1ml will be used fo half of the face.
  * After gentle cleansing, topical analgesic cream will be applied over the area to be treated.
  * The microneedles will be used, the skin will be stretched and microneedling will be carried out in vertical, horizontal, and both diagonal directions for about four to five times. Tranexamic acid, 0.5 to 1 ml (4 mg/mL), will be applied over this area, and the procedure will be repeated four to five times in the above-said directions
  Other Names: microneedling using tranxemic acid
  Arms: G II B (left side):will be treated by tranexemic acid

SUMMARY:
To compare the efficacy and safety of cryopeeling (using Liquid Nitrogen) and tranexemic acid (cyclokapron) versus chemical peeling (using TCA 20%) in treatment of melasma.

DETAILED DESCRIPTION:
Melasma is a common, acquired, circumscribed hypermelanosis of the sun-exposed skin, It presents as symmetric, hyperpigmented macules having irregular, serrated, and geographic borders , The most common locations are the cheeks, upper lips, the chin and the forehead, but other sun-exposed areas may also be occasionally involved .

Studies has indicated the role of several risk factors such as genetics, sunlight, age, gender, hormones, pregnancy, thyroid dysfunction, cosmetics and medications .

Histologic features of melasma include an increase in the content of both epidermal and dermal melanin, but the quantity varies with the intensity of hyperpigmentation. In addition, most studies show no quantitative increase in melanocytes; however, the cells are enlarged with prominent and elongated dendrites and more abundant melanosomes. Additional features of the involved skin include solar elastosis and increased mast cells, dermal blood vessels, and expression of vascular endothelial growth factor.

Commonly used topical agents for the treatment of melasma include hydroquinone, azelaic acid, kojic acid, glycolic acid, salicylic acid and tretinoin. Of these treatments, hydroquinone remains the gold standard .Second-line treatments, such as chemical peels and lasers, are efficacious in some patients .

Chemical peeling is the application of a chemical agent to the skin, which causes the controlled destruction of a part or of the entire epidermis with or without the dermis, leading to exfoliation and removal of superficial lesions, followed by regeneration of new epidermal and dermal tissues [khunger, 2008]. The mechanism of action in melasma is the removal of unwanted melanin via controlled chemical burn of the skin .

Trichloroacetic acid has been used as a peeling agent for a long time and is still the most effective and safest agent for medium peeling, Its depth of penetration depends on the TCA concentration and on the preparation of the skin, specially the degreasing. Between 10% and 30% concentration is considered a superficial peel; above 30% provides a medium-depth peel.

Cryopeeling is a technique that uses cryotherapy in a diffuse manner throughout the skin region affected by sun damage in order to promote cell renewal and desquamation, with possible benefits in the appearance of new lesions caused by photodamage. Up to the investigator's knowledge, few studies were performed evaluating such technique.

Recently, trans-4-(Aminomethyl) cyclohexanecarboxylic acid, or tranexamic acid (TA), has been proposed as a new treatment for melasma.The main mechanism of the hypopigmentant effects of TA is due to its antiplasmin activity .In addition, TA is similar to tyrosine in a portion of its structure, which can inhibit tyrosinase competitively .Also, Plasmin transforms the vascular endothelial growth factor (VEGF) into a diffusing form, and histological examination showed that TA plays an important role in the reduction of erythema and vascularities and the number of mast cell in the dermis.Various forms of TA are used orally, topically and as a microinjection for the treatment of melasma.

ELIGIBILITY:
Inclusion Criteria:

* -Subjects presented with melasma.
* Age 20-40 years old.
* Melasma persisting for more than 6 months that has failed to respond to conventional treatment with hydroquinone or other topical lightening agents.

Exclusion Criteria:

* -History of photosensitivity, keloids, hypertrophic scarring and post- inflammatory hyperpigmentation.
* Pregnancy and lactation.
* Subjects with local inflammatory skin disorder or active herpes infection at the site of procedure.
* Subjects with history of medical diseases which contraindicate cryosurgery such as; cold intolerance, cold urticaria, Raynaud's disease and history of allergic reactions to cryosurgery.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
melasma area and severity index (MASI) | baseline
  Clinical evaluation of melasma severity will be done by melasma area severity index (MASI) every session and at the end of treatment.
  No response, no improvement.
  * Mild response, <25% improvement.
  * Moderate response, 25% to < 50% improvement.
  * Good response, 50% to < 75% improvement.
  * Very good response, >75% improvement.
photo of the patient | baseline
  photo of the patient before and after treatment
Biopsy | baseline
  A punch biopsy will be taken from affected area for histipathological examination

REFERENCES:
- [Background] Kim EH, Kim YC, Lee ES, Kang HY. The vascular characteristics of melasma. J Dermatol Sci. 2007 May;46(2):111-6. doi: 10.1016/j.jdermsci.2007.01.009. Epub 2007 Mar 23. PMID 17363223
- [Background] Hexsel D, Rodrigues TC, Dal'Forno T, Zechmeister-Prado D, Lima MM. Melasma and pregnancy in southern Brazil. J Eur Acad Dermatol Venereol. 2009 Mar;23(3):367-8. doi: 10.1111/j.1468-3083.2008.02885.x. Epub 2008 Jul 7. No abstract available. PMID 18631207
- [Background] Sheth VM, Pandya AG. Melasma: a comprehensive update: part I. J Am Acad Dermatol. 2011 Oct;65(4):689-697. doi: 10.1016/j.jaad.2010.12.046. PMID 21920241
- [Background] Moin A, Jabery Z, Fallah N. Prevalence and awareness of melasma during pregnancy. Int J Dermatol. 2006 Mar;45(3):285-8. doi: 10.1111/j.1365-4632.2004.02470.x. PMID 16533230
- [Background] Sheth VM, Pandya AG. Melasma: a comprehensive update: part II. J Am Acad Dermatol. 2011 Oct;65(4):699-714. doi: 10.1016/j.jaad.2011.06.001. PMID 21920242
- [Background] Sarkar R, Bansal S, Garg VK. Chemical peels for melasma in dark-skinned patients. J Cutan Aesthet Surg. 2012 Oct;5(4):247-53. doi: 10.4103/0974-2077.104912. PMID 23378706
- [Background] Monheit GD, Chastain MA. Chemical peels. Facial Plast Surg Clin North Am. 2001 May;9(2):239-55, viii. PMID 11457690
- [Background] Perper M, Eber AE, Fayne R, Verne SH, Magno RJ, Cervantes J, ALharbi M, ALOmair I, Alfuraih A, Nouri K. Tranexamic Acid in the Treatment of Melasma: A Review of the Literature. Am J Clin Dermatol. 2017 Jun;18(3):373-381. doi: 10.1007/s40257-017-0263-3. PMID 28283893
- [Background] Na JI, Choi SY, Yang SH, Choi HR, Kang HY, Park KC. Effect of tranexamic acid on melasma: a clinical trial with histological evaluation. J Eur Acad Dermatol Venereol. 2013 Aug;27(8):1035-9. doi: 10.1111/j.1468-3083.2012.04464.x. Epub 2012 Feb 13. PMID 22329442
- [Background] Sharma YK, Gupta A. Some Other Serendipitous Discoveries in Dermatology. Indian J Dermatol. 2016 Jan-Feb;61(1):95-6. doi: 10.4103/0019-5154.174045. No abstract available. PMID 26955108